CLINICAL TRIAL: NCT06076642
Title: Long-term Safety and Tolerability of TAK-881 in Subjects With Primary Immunodeficiency Diseases (PIDD)
Brief Title: A Study About the Long-Term Safety of TAK-881 in People With Primary Immunodeficiency Diseases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Collaborators: Takeda Development Center Americas, Inc. (Industry); Baxalta Innovations GmbH, now part of Takeda (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAK-881-3002; 2023-505946-24-00 (EU CTIS Number)
Record Dates: First submitted 2023-10-04; First posted 2023-10-11 (Actual); Last update posted 2025-05-08 (Actual); Status verified 2025-05

CONDITIONS: Primary Immunodeficiency Diseases (PID)
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — gamma-Globulins; Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- TAK-881 (Experimental): Epoch 1: Participants who completed study TAK-881-3001 (NCT05755035) and met eligibility criteria will receive TAK-881 subcutaneous (SC) infusion using investigational needle sets at the same dose and same treatment interval as at the last infusion in TAK-881-3001 (NCT05755035) at Week 1 and at Weeks 13 and Week 25 of study TAK-881-3002.
  Epoch 2: Participants with anti-rHuPH20 antibody titer >=1:160 at any time point during Study TAK-881-3001 (NCT05755035) and/or Study TAK-881-3002 Epoch 1, will continue receiving TAK-881 every 12 weeks for up to Week 121.
  After the first TAK-881 infusion in study TAK-881-3002, the interval and/or the dose may be adjusted only at scheduled site visits at the investigator's discretion.
  Interventions: Biological: TAK-881; Device: SC Investigational Needle Sets

INTERVENTIONS:
Biological: TAK-881 — Participants will receive SC infusion of TAK-881.
  Other Names: Immune Globulin Subcutaneous (Human), 20% Solution with Recombinant Human Hyaluronidase (rHuPH20).
Device: SC Investigational Needle Sets — The single-use only SC needle set will be used to administer TAK-881 to the target depth below the skin surface. One needle set (single or bifurcated) will be used per infusion.

SUMMARY:
The main aim of this study is to learn if TAK-881 is safe and well tolerated during long-term use in adults and children with PIDD who are eligible and completed study TAK-881-3001 (NCT05755035).

The participants will receive the first dose of TAK-881 immunoglobulin (IgG) infusion at the same dosage as the last dose administered in study TAK-881-3001 (NCT05755035). After the first TAK-881 infusion in study TAK-881-3002, the dosing interval (can be adjusted by participant/caregiver) and/or the dose of TAK-881 can be adjusted by the study doctor to every 2, 3 or 4 weeks at scheduled site visits.

Participants will visit the clinic every 12 weeks until the End of Study (EOS) visit.

DETAILED DESCRIPTION:
The study consists of two Epochs: Epoch 1 and Epoch 2. In Epoch 1 eligible participants will have the opportunity to receive TAK-881 for a minimum of 6 months. After 6 months in study TAK-881-3002, the results of the anti-rHuPH20 binding antibody assay from either study TAK-881-3001 (NCT05755035) or study TAK-881-3002 (Epoch 1) will be used to determine the next steps in the study:

* Epoch 1: Participants with an anti-rHuPH20 antibody titer less than [<] 1:160 will complete the EOS visit on the day of the first non-investigational product (IP) infusion following Study Visit Week 25.
* Epoch 2: Participants with an anti-rHuPH20 antibody titer greater than or equal to [>=] 1:160 at any time point during Study TAK-881-3001 (NCT05755035) and/or study TAK-881-3002 (Epoch 1), will continue with an additional two years of TAK-881 treatment and undergo safety follow-up and will complete the EOS visit on the day of the first non-IP infusion following study Visit Week 121.

ELIGIBILITY:
Inclusion Criteria

Participants who meet ALL of the following criteria are eligible for this study:

* Participant must have completed Study TAK-881-3001 (NCT05755035).
* Participant/Participant's parent(s)/legal guardian(s) is/are willing and able to comply with the requirements of the protocol.
* Participant/Participant's parent(s)/legal guardian(s) has/have provided informed consent/assent (if applicable), including providing consent for use of the investigational medical device, prior to the initiation of any study procedures.

Exclusion Criteria

* Participant has a serious medical condition such that the participant's safety or medical care would be impacted by participation in this long-term follow-up study.
* New medical condition that developed during participation in Study TAK-881-3001 (NCT05755035), that, in the judgment of the investigator, could increase risk to the participant or interfere with the evaluation of TAK-881 and/or conduct of the study.
* Participant has participated in another clinical study involving an investigational product (IP) or investigational device within 30 days prior to screening (with the exception of Study TAK-881-3001 [NCT05755035]).
* Participant is scheduled to participate in another clinical study involving an IP or investigational device during the course of this study.
* Participant is a family member or employee of the investigator or the investigator's site staff.
* Women of childbearing potential who meet any one of the following criteria:-

  1. Participant has a positive pregnancy test.
  2. Participant does not agree to employ a highly effective form of contraception for the duration of the study.
* If female, participant is pregnant or lactating at the time of screening or intends to become pregnant or begin lactating during the study.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2024-11-04 (Actual); Primary Completion 2029-01-15 (Estimated); Study Completion 2029-01-15 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) | Up to Week 121
Number of Participants With Infusion Withdrawals, Interruptions, and Infusion Rate Reductions due to TAK-881-related TEAEs | Up to Week 121

SECONDARY OUTCOMES:
Annualized Rate of all Infections | Up to Week 121
Annualized Rate of Acute Serious Bacterial Infections (ASBIs) | Up to Week 121
Annualized Rate of Episodes of Fever | Up to Week 121
Time to First ASBI | Up to Week 121
Duration of Infections | Up to Week 121
Number of Participants With Positive Binding Antibodies and Neutralizing Antibodies to rHuPH20 | Up to Week 121
Trough Level of Total IgG | Up to Week 121
Doses of TAK-881 | Up to Week 121
Treatment Interval of TAK-881 | Up to Week 121
Number of Infusions Per Month With Investigational Medical Device Using TAK-881 | Up to Week 121
Number of Infusions Sites (Needle Sticks) per Month With Investigational Medical Device Using TAK-881 | Up to Week 121
Number of Infusions Sites (Needle Sticks) per infusion With Investigational Medical Device Using TAK-881 | Up to Week 121
Duration of Infusions (minutes) With Investigational Medical Device Using TAK-881 | Up to Week 121
Monthly Infusion Time (minutes/month) With Investigational Medical Device Using TAK-881 | Up to Week 121
Maximum Tolerated Infusion Rate per Site (milliliter/hour/site) With Investigational Medical Device Using TAK-881 | Up to Week 121
Infusion Volume per Site (milliliter/site) With Investigational Medical Device Using TAK-881 | Up to Week 121
Number of Participants who have Infusions of TAK-881 at Physical Location | Up to Week 121
  Physical location includes site/infusion center or home.
Number of Participants, Caregiver, or Healthcare Professional (HCP) who have Administration of TAK-881 | Up to Week 121
Treatment Satisfaction Questionnaire for Medication (TSQM-9) Scores in Participants Aged >=16 Years | From Week 13 up to Week 121
  TSQM-9 is a 9-item, validated, self-administered instrument to assess participants satisfaction with medication. It consists of 3 subscales: effectiveness, convenience and global satisfaction. The item scores of each of the 3 domains are summed and transformed to create a total score of 0 (extremely dissatisfied) to 100 (extremely satisfied). Higher score indicates greater satisfaction in that domain.
Health-Related Quality of Life (HRQoL): EuroQol 5 Dimension 5 Level Questionnaire (EQ-5D-5L) Score in Participants Aged >=12 Years | From Baseline up to Week 121
  The EQ-5D-5L is a validated, self-administered assessment of overall health designed by the EuroQol Group. The instrument consists of two components: the EQ-5D descriptive system and the standard vertical EQ visual analogue scale (EQ-VAS). The descriptive system consists of 5 dimensions (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression). Each dimension has five response categories: no problems, slight problems, some or moderate problems, severe problems, or extreme problems. Participants will be asked to describe their health state that day by choosing one of 5 responses that reflect the levels of severity for each of the 5 dimensions. The EQ-VAS measures one's self-perceived health today on a vertical scale from 0 (worst imaginable health) to 100 (best imaginable health) on which participants have to indicate their current health. Higher score indicates best health status.
Treatment Preference Measured by a Disease-specific Questionnaire for Participants and the Investigational Medical Device Using TAK-881 in Participants Aged >=12 Years | At Weeks 25 and 73
  The disease-specific treatment preference questionnaire is a self-administered, non-validated scale to assess participant preference for various attributes of IgG therapy and accompanying devices, such as ease of use of administration of TAK-881 complexity of administration, and convenience. The questionnaire consists of two components. The first component asks participants to indicate the extent to which they like or dislike aspects of TAK-881, including treatment frequency, time, ease, convenience, and complexity. Each item has five response categories: like very much, like, no preference, dislike, and dislike very much. The second component is a single question asking whether they would choose to continue receiving treatment after the trial ends.
Number of Days not Able to go to School, Work, Daycare, or to Perform Normal Daily Activities Due to Infections and/or their Treatment or Other Illnesses | Up to Week 121
Number of Days on Antibiotics | Up to Week 121
Number of Hospitalizations With Indications (Infection or other Illnesses) | Up to Week 121
Number of Days of Hospitalization | Up to Week 121
Number of Acute Physician Visits Due to Infection or Other Illnesses | Up to Week 121
Infusion Preparation Time For TAK-881 by HCP | Up to Week 121
Infusion Preparation Time For TAK-881 by Participants/Caregiver | Up to Week 121
Number of Participants With Adverse Events (AEs) Related to the Investigational Medical Device | Up to Week 121

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (5):
- United States (5):
  - Central Georgia Infectious Disease Consultants, Macon, Georgia
  - Sneeze, Wheeze, & Itch Associates, LLC, Normal, Illinois
  - Montefiore Medical Center, The Bronx, New York
  - Duke Asthma, Allergy and Airway Center, Durham, North Carolina
  - Allergy Partners of North Texas, Dallas, Texas

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/11d16226ed664112?idFilter=%5B%22TAK-881-3002%22%5D